CLINICAL TRIAL: NCT04107116
Title: Enhancing Community Capacity to Improve Cancer Care Delivery: The Effect of a Lay Health Worker Intervention on Patient-reported Symptoms, Healthcare Use, Total Costs of Care, and End-of-life Care Delivery
Brief Title: Enhancing Community Capacity to Improve Cancer Care Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 455
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: End of Life; Cancer
Keywords: cancer end of life patient-centered
MeSH Terms: conditions — Death; Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group Arm (Experimental): Patients randomized into the intervention will be assigned a lay health worker who will contact the patient to begin the intervention. The intervention includes: proactive symptom assessments for patients for up to 12-months.
  Interventions: Behavioral: Program participants; Other: Usual Care
- Control Group Arm (Active Comparator): The control group arm will receive usual care as provided by their local oncologists.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Program participants — The intervention is a 12-month telephonic program in which a lay health worker (LHW), supervised on-site by a registered nurse practitioner (RNP), assessed patient symptoms after diagnosis using the validated Edmonton Symptom Assessment Scale (ESAS) (cite) with the frequency of symptom assessment varying based on patient risk.
  Arms: Intervention Group Arm
Other: Usual Care — Usual care as provided by local oncologists

SUMMARY:
Undertreated patient symptoms and resulting acute care use require approaches that improve symptom-burden. Previously a a lay health worker (LHW)-led symptom screening intervention was developed for patients with advanced cancer. This intervention will be expanded to all patients with cancer and the LHW will be trained to refer patients to palliative care and behavioral health. This intervention will evaluate the effect on symptom-burden, survival, healthcare use, and total costs.

DETAILED DESCRIPTION:
From 11/1/2016 - 9/30/2018, all newly diagnosed Medicare Advantage enrollees with solid or hematologic malignancies were enrolled in the intervention. Outcomes were compared outcomes to patients in the year prior (control arm). The primary outcome was change in symptoms using the Edmonton Symptom Assessment Scale (ESAS) and Personal Health Questionnaire-9 (PHQ-9) at baseline, 6- and 12-months post-enrollment. Secondary outcomes were between-group comparison of survival, 12-month healthcare use and costs.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with cancer
* Diagnosis of relapse or progressive disease (any cancer diagnosis) as identified by imaging or biopsy and confirmed by physician.
* Must be 18 years or older.
* Must have capacity to verbally consent

Exclusion Criteria:

-Inability to consent to the study due to lack of capacity as documented by the referring physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manali I Patel, MD MPH MS, Principal Investigator — Stanford University
Locations (1):
- Oncology Institute for Hope and Innovation, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted with participants care for in 9 of 10 oncology clinics within the Oncology Institute of Hope and Innovation. Participants were screened by a new patient coordinator, then enrolled from 11/1/2016 to 10/31/2017 and were followed up with for 12 months after or death.
Pre-assignment Details: One oncology clinic was excluded due to involvement in a previously reported intervention in the sources. The study also excluded clinic patients that did not receive medical oncology care.
Period: Overall Study
Arm/Group | Intervention Group Arm | Control Group Arm
Started | 425 | 407
Completed | 425 | 407
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Amongst the 832 participants, 6 baseline characteristics were measured between the intervention and control arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group Arm | Control Group Arm | Total
Number analyzed (Participants) | 425 | 407 | 832
Age, Customized [Mean (Standard Deviation); unit: years] — Population: The total participant population was broken down into each of the 9 individual clinic sites, and then analyzed.
  years
    Clinic A: number analyzed (Participants) | 80 | 75 | 155
    Clinic A | 79.6 (10.2) | 78.6 (10.3) | 79.2 (10.2)
    Clinic B: number analyzed (Participants) | 47 | 45 | 92
    Clinic B | 79.5 (9.8) | 79.3 (9.1) | 79.4 (9.3)
    Clinic C: number analyzed (Participants) | 44 | 42 | 86
    Clinic C | 78.1 (10.2) | 80.0 (10.6) | 79.2 (10.8)
    Clinic D: number analyzed (Participants) | 39 | 39 | 78
    Clinic D | 77.1 (10.2) | 80.0 (11.2) | 78 (10.9)
    Clinic E: number analyzed (Participants) | 45 | 44 | 89
    Clinic E | 78.9 (10.4) | 80.7 (10.2) | 79 (10.3)
    Clinic F: number analyzed (Participants) | 42 | 40 | 82
    Clinic F | 80.0 (10.2) | 79.4 (10.3) | 79.8 (10.2)
    Clinic G: number analyzed (Participants) | 40 | 38 | 78
    Clinic G | 77.5 (10.4) | 77.7 (10.2) | 77.6 (10.2)
    Clinic H: number analyzed (Participants) | 47 | 43 | 90
    Clinic H | 76.4 (10.1) | 77.9 (10.2) | 76.8 (10.1)
    Clinic I: number analyzed (Participants) | 41 | 41 | 82
    Clinic I | 77.2 (10.2) | 78.9 (10.1) | 78 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The total participant population was broken down into each of the 9 individual clinic sites, and then analyzed.
  Participants
    Clinic A: number analyzed (Participants) | 80 | 75 | 155
    Clinic A: Female | 38 | 25 | 63
    Clinic A: Male | 42 | 50 | 92
    Clinic B: number analyzed (Participants) | 47 | 45 | 92
    Clinic B: Female | 23 | 17 | 40
    Clinic B: Male | 24 | 28 | 52
    Clinic C: number analyzed (Participants) | 44 | 42 | 86
    Clinic C: Female | 20 | 12 | 32
    Clinic C: Male | 24 | 30 | 54
    Clinic D: number analyzed (Participants) | 39 | 39 | 78
    Clinic D: Female | 12 | 18 | 30
    Clinic D: Male | 27 | 21 | 48
    Clinic E: number analyzed (Participants) | 45 | 44 | 89
    Clinic E: Female | 20 | 16 | 36
    Clinic E: Male | 25 | 28 | 53
    Clinic F: number analyzed (Participants) | 42 | 40 | 82
    Clinic F: Female | 20 | 19 | 39
    Clinic F: Male | 22 | 21 | 43
    Clinic G: number analyzed (Participants) | 40 | 38 | 78
    Clinic G: Female | 15 | 21 | 36
    Clinic G: Male | 25 | 17 | 42
    Clinic H: number analyzed (Participants) | 47 | 43 | 90
    Clinic H: Female | 23 | 13 | 36
    Clinic H: Male | 24 | 30 | 54
    Clinic I: number analyzed (Participants) | 41 | 41 | 82
    Clinic I: Female | 20 | 13 | 33
    Clinic I: Male | 21 | 28 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The total participant population was broken down into each of the 9 individual clinic sites, and then analyzed.
  Participants
    Clinic A: number analyzed (Participants) | 80 | 75 | 155
    Clinic A: Non-Hispanic White | 38 | 36 | 74
    Clinic A: Hispanic | 37 | 28 | 65
    Clinic A: Non-Hispanic Black | 3 | 6 | 9
    Clinic A: Asian Pacific Islander | 1 | 3 | 4
    Clinic A: Native Hawaiian, Alaskan Native, or American Indian | 1 | 2 | 3
    Clinic B: number analyzed (Participants) | 47 | 45 | 92
    Clinic B: Non-Hispanic White | 25 | 18 | 43
    Clinic B: Hispanic | 18 | 21 | 39
    Clinic B: Non-Hispanic Black | 3 | 3 | 6
    Clinic B: Asian Pacific Islander | 1 | 1 | 2
    Clinic B: Native Hawaiian, Alaskan Native, or American Indian | 0 | 2 | 2
    Clinic C: number analyzed (Participants) | 44 | 42 | 86
    Clinic C: Non-Hispanic White | 25 | 22 | 47
    Clinic C: Hispanic | 17 | 17 | 34
    Clinic C: Non-Hispanic Black | 1 | 1 | 2
    Clinic C: Asian Pacific Islander | 1 | 2 | 3
    Clinic C: Native Hawaiian, Alaskan Native, or American Indian | 0 | 0 | 0
    Clinic D: number analyzed (Participants) | 39 | 39 | 78
    Clinic D: Non-Hispanic White | 16 | 20 | 36
    Clinic D: Hispanic | 20 | 15 | 35
    Clinic D: Non-Hispanic Black | 1 | 1 | 2
    Clinic D: Asian Pacific Islander | 2 | 2 | 4
    Clinic D: Native Hawaiian, Alaskan Native, or American Indian | 0 | 1 | 1
    Clinic E: number analyzed (Participants) | 45 | 44 | 89
    Clinic E: Non-Hispanic White | 18 | 15 | 33
    Clinic E: Hispanic | 19 | 24 | 43
    Clinic E: Non-Hispanic Black | 1 | 2 | 3
    Clinic E: Asian Pacific Islander | 3 | 3 | 6
    Clinic E: Native Hawaiian, Alaskan Native, or American Indian | 4 | 0 | 4
    Clinic F: number analyzed (Participants) | 42 | 40 | 82
    Clinic F: Non-Hispanic White | 20 | 23 | 43
    Clinic F: Hispanic | 21 | 11 | 32
    Clinic F: Non-Hispanic Black | 1 | 1 | 2
    Clinic F: Asian Pacific Islander | 0 | 3 | 3
    Clinic F: Native Hawaiian, Alaskan Native, or American Indian | 0 | 2 | 2
    Clinic G: number analyzed (Participants) | 40 | 38 | 78
    Clinic G: Non-Hispanic White | 21 | 22 | 43
    Clinic G: Hispanic | 19 | 12 | 31
    Clinic G: Non-Hispanic Black | 0 | 0 | 0
    Clinic G: Asian Pacific Islander | 0 | 2 | 2
    Clinic G: Native Hawaiian, Alaskan Native, or American Indian | 0 | 2 | 2
    Clinic H: number analyzed (Participants) | 47 | 43 | 90
    Clinic H: Non-Hispanic White | 22 | 21 | 43
    Clinic H: Hispanic | 21 | 17 | 38
    Clinic H: Non-Hispanic Black | 0 | 1 | 1
    Clinic H: Asian Pacific Islander | 0 | 2 | 2
    Clinic H: Native Hawaiian, Alaskan Native, or American Indian | 4 | 2 | 6
    Clinic I: number analyzed (Participants) | 41 | 41 | 82
    Clinic I: Non-Hispanic White | 23 | 22 | 45
    Clinic I: Hispanic | 14 | 16 | 30
    Clinic I: Non-Hispanic Black | 1 | 1 | 2
    Clinic I: Asian Pacific Islander | 2 | 2 | 4
    Clinic I: Native Hawaiian, Alaskan Native, or American Indian | 1 | 0 | 1
Cancer diagnosis [Count of Participants; unit: Participants] — Population: The total participant population was broken down into each of the 9 individual clinic sites, and then analyzed.
  Participants
    Clinic A: number analyzed (Participants) | 80 | 75 | 155
    Clinic A: Thoracic | 8 | 6 | 14
    Clinic A: Gastrointestinal | 19 | 19 | 38
    Clinic A: Head and neck | 4 | 3 | 7
    Clinic A: Malignant hematologic | 4 | 6 | 10
    Clinic A: Genitourinary | 17 | 8 | 25
    Clinic A: Other (skin, brain, bone, soft tissue, or head and neck) | 9 | 9 | 18
    Clinic A: Breast | 19 | 24 | 43
    Clinic B: number analyzed (Participants) | 47 | 45 | 92
    Clinic B: Thoracic | 7 | 5 | 12
    Clinic B: Gastrointestinal | 10 | 12 | 22
    Clinic B: Head and neck | 3 | 2 | 5
    Clinic B: Malignant hematologic | 7 | 6 | 13
    Clinic B: Genitourinary | 4 | 4 | 8
    Clinic B: Other (skin, brain, bone, soft tissue, or head and neck) | 6 | 7 | 13
    Clinic B: Breast | 10 | 9 | 19
    Clinic C: number analyzed (Participants) | 44 | 42 | 86
    Clinic C: Thoracic | 4 | 4 | 8
    Clinic C: Gastrointestinal | 7 | 9 | 16
    Clinic C: Head and neck | 1 | 0 | 1
    Clinic C: Malignant hematologic | 4 | 7 | 11
    Clinic C: Genitourinary | 5 | 4 | 9
    Clinic C: Other (skin, brain, bone, soft tissue, or head and neck) | 8 | 4 | 12
    Clinic C: Breast | 15 | 14 | 29
    Clinic D: number analyzed (Participants) | 39 | 39 | 78
    Clinic D: Thoracic | 5 | 4 | 9
    Clinic D: Gastrointestinal | 10 | 11 | 21
    Clinic D: Head and neck | 0 | 1 | 1
    Clinic D: Malignant hematologic | 1 | 4 | 5
    Clinic D: Genitourinary | 3 | 8 | 11
    Clinic D: Other (skin, brain, bone, soft tissue, or head and neck) | 7 | 2 | 9
    Clinic D: Breast | 13 | 9 | 22
    Clinic E: number analyzed (Participants) | 45 | 44 | 89
    Clinic E: Thoracic | 1 | 5 | 6
    Clinic E: Gastrointestinal | 15 | 10 | 25
    Clinic E: Head and neck | 1 | 2 | 3
    Clinic E: Malignant hematologic | 5 | 6 | 11
    Clinic E: Genitourinary | 9 | 4 | 13
    Clinic E: Other (skin, brain, bone, soft tissue, or head and neck) | 8 | 3 | 11
    Clinic E: Breast | 6 | 14 | 20
    Clinic F: number analyzed (Participants) | 42 | 40 | 82
    Clinic F: Thoracic | 7 | 3 | 10
    Clinic F: Gastrointestinal | 10 | 13 | 23
    Clinic F: Head and neck | 2 | 1 | 3
    Clinic F: Malignant hematologic | 4 | 3 | 7
    Clinic F: Genitourinary | 4 | 5 | 9
    Clinic F: Other (skin, brain, bone, soft tissue, or head and neck) | 5 | 3 | 8
    Clinic F: Breast | 10 | 12 | 22
    Clinic G: number analyzed (Participants) | 40 | 38 | 78
    Clinic G: Thoracic | 3 | 3 | 6
    Clinic G: Gastrointestinal | 16 | 13 | 29
    Clinic G: Head and neck | 0 | 0 | 0
    Clinic G: Malignant hematologic | 4 | 5 | 9
    Clinic G: Genitourinary | 6 | 7 | 13
    Clinic G: Other (skin, brain, bone, soft tissue, or head and neck) | 3 | 2 | 5
    Clinic G: Breast | 8 | 8 | 16
    Clinic H: number analyzed (Participants) | 47 | 43 | 90
    Clinic H: Thoracic | 3 | 3 | 6
    Clinic H: Gastrointestinal | 20 | 16 | 36
    Clinic H: Head and neck | 3 | 0 | 3
    Clinic H: Malignant hematologic | 8 | 4 | 12
    Clinic H: Genitourinary | 3 | 1 | 4
    Clinic H: Other (skin, brain, bone, soft tissue, or head and neck) | 2 | 4 | 6
    Clinic H: Breast | 8 | 15 | 23
    Clinic I: number analyzed (Participants) | 41 | 41 | 82
    Clinic I: Thoracic | 5 | 6 | 11
    Clinic I: Gastrointestinal | 10 | 13 | 23
    Clinic I: Head and neck | 3 | 1 | 4
    Clinic I: Malignant hematologic | 5 | 4 | 9
    Clinic I: Genitourinary | 6 | 1 | 7
    Clinic I: Other (skin, brain, bone, soft tissue, or head and neck) | 7 | 4 | 11
    Clinic I: Breast | 5 | 12 | 17
Cancer Stage [Count of Participants; unit: Participants] — Cancer stages: stage 0 - the cancer is where it started (in situ) and hasn't spread; stage 1 - the cancer is small and hasn't spread anywhere else; stage 2 - the cancer has grown, but hasn't spread; stage 3 - the cancer is larger and may have spread to the surrounding tissues and/or the lymph nodes (or "glands", part of the immune system); stage 4 - the cancer has spread from where it started to at least 1 other body organ, also known as "secondary" or "metastatic" cancer. Stage was abstracted through chart review of clinical notes documented in the electronic health record by the oncologist. Population: The total participant population was broken down into each of the 9 individual clinic sites, and then analyzed.
  Participants
    Clinic A: number analyzed (Participants) | 80 | 75 | 155
    Clinic A: I | 14 | 13 | 27
    Clinic A: II | 16 | 16 | 32
    Clinic A: III | 18 | 12 | 30
    Clinic A: IV | 32 | 34 | 66
    Clinic B: number analyzed (Participants) | 47 | 45 | 92
    Clinic B: I | 11 | 14 | 25
    Clinic B: II | 9 | 5 | 14
    Clinic B: III | 9 | 4 | 13
    Clinic B: IV | 18 | 22 | 40
    Clinic C: number analyzed (Participants) | 44 | 42 | 86
    Clinic C: I | 13 | 13 | 26
    Clinic C: II | 11 | 6 | 17
    Clinic C: III | 6 | 7 | 13
    Clinic C: IV | 14 | 16 | 30
    Clinic D: number analyzed (Participants) | 39 | 39 | 78
    Clinic D: I | 7 | 5 | 12
    Clinic D: II | 6 | 8 | 14
    Clinic D: III | 11 | 11 | 22
    Clinic D: IV | 15 | 15 | 30
    Clinic E: number analyzed (Participants) | 49 | 44 | 93
    Clinic E: I | 9 | 9 | 18
    Clinic E: II | 8 | 8 | 16
    Clinic E: III | 10 | 8 | 18
    Clinic E: IV | 22 | 19 | 41
    Clinic F: number analyzed (Participants) | 42 | 40 | 82
    Clinic F: I | 11 | 12 | 23
    Clinic F: II | 7 | 7 | 14
    Clinic F: III | 5 | 6 | 11
    Clinic F: IV | 19 | 15 | 34
    Clinic G: number analyzed (Participants) | 40 | 38 | 78
    Clinic G: I | 10 | 5 | 15
    Clinic G: II | 5 | 5 | 10
    Clinic G: III | 9 | 7 | 16
    Clinic G: IV | 16 | 21 | 37
    Clinic H: number analyzed (Participants) | 47 | 43 | 90
    Clinic H: I | 12 | 11 | 23
    Clinic H: II | 10 | 9 | 19
    Clinic H: III | 7 | 6 | 13
    Clinic H: IV | 18 | 17 | 35
    Clinic I: number analyzed (Participants) | 41 | 41 | 82
    Clinic I: I | 5 | 9 | 14
    Clinic I: II | 11 | 5 | 16
    Clinic I: III | 6 | 8 | 14
    Clinic I: IV | 19 | 19 | 38
Risk Adjustment Factor [Mean (Standard Deviation); unit: Risk Adjustment Factor Score] — Risk Adjustment Factor (RAF) score range from 0 to no maximum value. Scores above 1.0 are considered high risk: RAF score range: RAF scores typically range from 0.6 to 1.2. A score of 1.0 is average, with decimal places representing percentages above or below average. A score above 1.0 indicates a higher risk of illness, while a score below 1.0 indicates a lower risk.RAF scores are used to calculate payments to healthcare organizations. RAF scores are based on a patient's disease burden and demographic information, adjusted for age, sex, and regionally based on costs of care. Population: The total participant population was broken down into each of the 9 individual clinic sites, and then analyzed.
  Risk Adjustment Factor Score
    Clinic A: number analyzed (Participants) | 80 | 75 | 155
    Clinic A | 2.96 (1.86) | 2.69 (1.86) | 2.88 (1.86)
    Clinic B: number analyzed (Participants) | 47 | 45 | 92
    Clinic B | 2.54 (1.37) | 2.89 (2.08) | 2.76 (1.88)
    Clinic C: number analyzed (Participants) | 44 | 42 | 86
    Clinic C | 2.23 (1.65) | 2.67 (1.70) | 2.43 (1.66)
    Clinic D: number analyzed (Participants) | 39 | 39 | 78
    Clinic D | 2.42 (1.69) | 2.69 (1.74) | 2.52 (1.71)
    Clinic E: number analyzed (Participants) | 45 | 44 | 89
    Clinic E | 2.59 (1.75) | 2.55 (1.99) | 2.56 (1.88)
    Clinic F: number analyzed (Participants) | 42 | 40 | 82
    Clinic F | 2.22 (1.82) | 2.76 (1.66) | 2.44 (1.72)
    Clinic G: number analyzed (Participants) | 40 | 38 | 78
    Clinic G | 2.84 (2.07) | 2.56 (1.73) | 2.67 (1.89)
    Clinic H: number analyzed (Participants) | 47 | 43 | 90
    Clinic H | 2.73 (2.12) | 2.46 (1.22) | 2.52 (1.82)
    Clinic I: number analyzed (Participants) | 41 | 41 | 82
    Clinic I | 2.93 (1.79) | 2.83 (2.23) | 2.87 (2.11)

OUTCOME MEASURES:

1. Primary Outcome: Edmonton Symptom Assessment Scale (ESAS) Symptom Screen
Description: Each patient will receive a quantitative symptom assessment survey (Edmonton Symptom Assessment Scale). Participants rate the intensity of 10 symptoms, each on a 11-point scale (0 to 10); sub-scores are then summed and averaged to create a total symptom score (range: 0 to 10, with 10 corresponding to worst symptom severity).
Time Frame: Baseline (at time of patient enrollment)
Measure: Mean (Full Range); unit: total score on a scale
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
total score on a scale | 7 [0 to 10] | 7 [0 to 10]

2. Primary Outcome: Edmonton Symptom Assessment Scale (ESAS) Symptom Screen
Description: as for outcome 1
Time Frame: 6 months after patient enrollment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 367 | 336
score on a scale | 8.2 [0 to 9] | 9.8 [5 to 10]

3. Primary Outcome: Edmonton Symptom Assessment Scale (ESAS) Symptom Screen
Description: as for outcome 1
Time Frame: 12 months after patient enrollment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 245 | 218
score on a scale | 7 [0 to 7] | 9.8 [6 to 10]

4. Primary Outcome: Personal Health Questionnaire-9 (PHQ-9) Depression Screen
Description: Each patient will receive a Personal Health Questionnaire-9 (PHQ-9) at baseline. PHQ-9 is measured on a scale of 0-27, where scores of 5, 10, 15, and 20 are cut-points for mild, moderate, moderately severe and severe depression, respectively.
Time Frame: Baseline (at time of patient enrollment)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
units on a scale | 2.9 [0 to 27] | 2.7 [0 to 27]

5. Primary Outcome: Personal Health Questionnaire-9 (PHQ-9) Depression Screen
Description: Each patient will receive a Personal Health Questionnaire-9 (PHQ-9) at 6 months. PHQ-9 is measured on a scale of 0-27, where scores of 5, 10, 15, and 20 are cut-points for mild, moderate, moderately severe and severe depression, respectively.
Time Frame: 6 months after patient enrollment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 367 | 336
score on a scale | 2.5 [0 to 27] | 2.9 [0 to 27]

6. Primary Outcome: Personal Health Questionnaire-9 (PHQ-9) Depression Screen
Description: Each patient will receive a Personal Health Questionnaire-9 (PHQ-9) at 12 months. PHQ-9 is measured on a scale of 0-27, where scores of 5, 10, 15, and 20 are cut-points for mild, moderate, moderately severe and severe depression, respectively.
Time Frame: 12 months after patient enrollment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 245 | 218
score on a scale | 1.9 [0 to 27] | 3.9 [0 to 27]

7. Secondary Outcome: Incidence of Emergency Department Visits Within 12-months After Patient Enrollment (Chart Review)
Description: Emergency Department use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment. We will evaluate comparisons of the number of visits (per 1000 members/year) with emergency department visits between study arms.
Time Frame: 12 months after patient enrollment
Measure: Number; unit: visits per 1000 members/yr.
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
visits per 1000 members/yr. | 0.43 | 0.57

8. Secondary Outcome: Incidence of Hospitalization Visits Within 12 Months After Patient Enrollment (Chart Review)
Description: Hospital use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment. We will evaluate comparisons of the number of visits (per 1000 members/year) with hospital use between study arms.
Time Frame: 12 months after patient enrollment
Measure: Number; unit: visits per 1000 members/yr.
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
visits per 1000 members/yr. | 0.54 | 0.72

9. Secondary Outcome: Number of Patients With a Hospice Consult Within 12-months After Patient Enrollment (Chart Review)
Description: Hospice consult for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
Participants | 207 | 101

10. Secondary Outcome: Total Health Care Costs (Claims Review)
Description: Total Health Care Costs for each patient will be abstracted by medical claims data review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Median (Inter-Quartile Range); unit: $USD
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
$USD | 17,869 [6,865 to 32,540] | 18,473 [6,415 to 37,910]

11. Secondary Outcome: Number of Patients With an Acute Care Facility Death (Chart Review)
Description: Acute Care Facility Deaths for each patient will be abstracted by electronic medical record chart review and claims review for each patient who has died at 12-months followup. We will evaluate comparisons of Acute Care Facility Deaths between study arms.
Time Frame: 30 days prior to death for patients who died at 12-months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
Participants | 18 | 30

12. Secondary Outcome: Number of Emergency Department Visit in the Last 30 Days of Life (Chart Review)
Description: Emergency Department (acute care) use for each patient will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of emergency department visits between study arms.
Time Frame: 30 days prior to death for patients who died at 12-months follow-up
Measure: Mean (Standard Deviation); unit: acute care visits
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
acute care visits | 0.10 (0.30) | 0.30 (0.46)

13. Secondary Outcome: Number of Hospitalization Visits in the Last 30 Days of Life (Chart Review)
Description: Hospital use for each patient will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of hospitalization use between study arms.
Time Frame: 30 days prior to death for patients who died at 12-months follow-up
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
hospitalizations | 0.27 (0.44) | 0.43 (0.82)

14. Secondary Outcome: Number of Patients With a Hospice Consult in the Last 30 Days of Life (Chart Review)
Description: Hospice use for each patient will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of hospice use between study arms.
Time Frame: 30 days prior to death for patients who died at 12-months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
Participants | 125 | 79

15. Secondary Outcome: Total Costs of Care (Claims Review)
Description: Total costs of care for each patient will be obtained through claims data for each patient for each patient who has died. We will evaluate comparisons of Total costs of care between study arms.
Time Frame: 30 days prior to death for patients who died at 12-months follow-up
Measure: Median (Inter-Quartile Range); unit: $USD
Arm/Group | Intervention Group Arm | Control Group Arm
Number analyzed (Participants) | 425 | 407
$USD | 3,602 [1,076 to 9,436] | 12,726 [5,259 to 22,170]

ADVERSE EVENTS:
Time Frame: The time frame over which the adverse data were collected were from time of enrollment until 1 year after enrollment.
Arm/Group | Intervention Group Arm | Control Group Arm
All-Cause Mortality (participants affected / at risk) | 180/425 | 189/407
Serious Adverse Events (participants affected / at risk) | 0/425 | 0/407
Other Adverse Events (participants affected / at risk) | 0/425 | 0/407

LIMITATIONS AND CAVEATS:
Patients in the intervention group were compared with a retrospective cohort of patients; the practice setting was limited to 9 clinics associated with one institution; there may be differences in unmeasured variables, which would bias the findings; could not measure the physician assistant interventions made in response to symptoms. Could not assess the result of the intervention on intermediary variables due to only collecting data on palliative care and behavioral health.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT04107116/Prot_000.pdf